CLINICAL TRIAL: NCT04074239
Title: Using Video Transmission for Optimized Telephone Triage of Children With Fever at the Medical Helpline 1813 in Copenhagen, Denmark
Brief Title: Using Video for Triage of Children With Fever at the Medical Helpline 1813 in Copenhagen, Denmark
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Copenhagen University Hospital at Herlev (Other); Rigshospitalet, Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Video fever
Record Dates: First submitted 2019-08-14; First posted 2019-08-30 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Fever; Telemedicine; Pediatrics; Triage
Keywords: telemedicine; Triage; Call centers; Fever; Pediatrics
MeSH Terms: conditions — Fever

STUDY DESIGN:
Intervention Model Description: The operators at the medical helpline 1813 will triage children meeting the inclusion criteria by video every other day they are at work, and by telephone the other days. The children will hence be randomized to either video or telephone depending on what day they are calling and which operator they are talking to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video triage (Experimental): The sick child will be triaged on video by the operator.
  Interventions: Other: Video triage
- Telephone triage (No Intervention): The sick child will be triaged solely on telephone by the operator.

INTERVENTIONS:
Other: Video triage — The operator at the Medical Helpline will offer the parent who's calling regarding the sick child to assess the child on video, as compared to the routine way; on the telephone.
  Arms: Video triage

SUMMARY:
Background:

The Medical Helpline 1813 in Copenhagen, Denmark handles acute, non-life threatening medical emergencies. Approx. 200,000 calls/year concern children, and about 30% are referred to a pediatric urgent care center. However, most of these children have very mild symptoms, which require neither treatment nor tests, merely parental guidance.

Initial assessment; triage, of children on the phone is difficult, especially when the operator does not know the child or family, and when it is difficult to describe the symptoms in medical terms. This may result in too many not-so-sick children and too few more severely sick children getting sent to hospital.

Many parents are very worried about their sick child, but it is not known if this worry can be integrated in the triage process.

Purpose:

It will be studied if triage by video calls; video triage; provide greater security for parents and call operators so that more children can stay at home after medical guidance, causing at least 10% fewer visits to pediatric urgent care centers. The degree of worry of the parents will also be registered.

Method:

Children aged 3 months to 5 years with fever will be triaged by either video or telephone every other day, to compare the results between these to otherwise similar groups. Operators and parents answer surveys about their experiences.

Yield:

Video triage can "give eyes to the operators" and revolutionize telephone triage. The study may result in fewer children referred to hospitals, more appropriate use of resources and better experiences for the families.

DETAILED DESCRIPTION:
Background Each year, the Copenhagen Emergency Services receives approx. 190,000 calls to the Medical Helpline 1813 regarding sick children younger than 12 years (injuries excluded). These children are not so sick that the parents call 112, but the parents need to get in contact with the health services outside their general practitioners' (GP) opening hours.

The health professionals at 1813, have several options after the conversation with the parent. They can for example admit the children at a Pediatric Emergency Department (PED), refer them to assessment in a pediatric urgency care clinic (Børnelægevagten), guide the parents in care for the child (self-care), or advise them to see their GP the next working day. Of the 190,000 calls annually regarding sick children, the majority is concerning young children; in 2018, just over 175,000 of the calls concerned children under the age of 6. Approx. 30% of these children were referred to assessment in a pediatric urgency care clinic. Most of these children reveal to have quite mild symptoms, and most are sent back home with good advice after an assessment by a doctor.

Phone triage is difficult, especially when the operator does not know the child nor the parents, and it may be difficult to describe symptoms with words. Many visits to the pediatric urgency care clinic can be perceived as unnecessary and inappropriate for the sick child and its parents, whom, with advice and proper guidance could have stayed at home. Moreover, the visits are expensive for the health system.

A Danish study, which was conducted the first year after the 1813 helpline was launched, showed that most calls concerned children aged 0-1 years and that the calls seldom were about serious conditions. The author interpreted the results as if the parents were primarily calling 1813 to feel safe about the child's condition.

In a Danish study from 2013, 28% of the urgent inquiries outside the GP's opening hours concerned just 2.5% of the children. These children had at least 4 of such urgent inquiries in one year. The median age of these children was 2.9 years old, as compared to 7.3 years in the whole group of children. The five most common working diagnoses among the children with many contacts were acute bronchitis, viral disease, seizures (not classified elsewhere), abdominal pain and gastroenteritis, that is, conditions where children are likely to have a fever. The authors mention that fever in itself causes many contacts to the health services and that the parents are very concerned about fever, which is also shown in several international studies.

It is recommended that all febrile children younger than the age of 3 months shall be seen by a doctor urgently. This is due to it being difficult to assess so young children and that such young children are likely to have a serious infectious disease. The initial assessment of the older febrile children can also be difficult. A study conducted in Belgian GPs involving 4,000 children with acute disease showed that only 0.8% of children had a serious infectious disease demanding hospitalization. The doctor's feeling that "something is wrong" was the most important factor in identifying these seriously ill children during the initial medical consultation. The authors then developed a "five step decision tree", where "something is wrong" is the first step. The tool has proven to provide the best results in terms of diagnostic safety in a validation study. The low incidence of severe infectious diseases in industrialized countries has also been shown in other studies.

In 2017, a novel scale grading the worry of patients was developed in a Ph.D. project at 1813. It is called degree-of-worry (DOW). The patients scored their worry from 1-5, with 1 being minimally worried and 5 being maximally worried, and it was subsequently studied if the DOW could predict the risk of the patients being hospitalized. The question of if DOW also can be used by parents calling 1813 about their sick child is not yet answered.

Telemedicine is gaining greater and greater acceptance in the medical world, also within pediatrics. The American Academy of Pediatrics has urged both general pediatricians and pediatric subspecialists to use telemedicine to be able to help more children. In Denmark, there are also several initiatives within telemedicine regarding adults. While these initiatives are being introduced, it must be remembered that there is a limited amount of evidence-based knowledge about the use of video in the health care field, not least in the field of triage.

An American study examined if febrile children could be evaluated on video using the Yale Observation Scale. The Yale Observation Scale is an assessment tool designed to predict serious illness in febrile children. The American scientists filmed febrile children in a Pediatric Emergency Department and found that assessment by the Yale Observation Scale of the children on film corresponded to the assessment made by the doctors who conducted a regular bedside examination.

The project group launched a video triage project at 1813 earlier in 2019, using video in calls regarding children with respiratory symptoms. The initial results show that the setup works and that there is a high level of satisfaction in both parents and operators. This project concerning febrile children is analog to the latter project, only with minor changes and also with a new focus on the degree of worry.

Purpose It will be investigated if video calls using the parents' smartphones can improve the assessment of febrile children when contacting the Medical Helpline 1813. The hypothesis is that video calls can optimize the referral within the next 8 hours after the call, so that more parents can feel safe staying home with their only slightly ill child, and that more children with severe symptoms are referred directly to admission at a Pediatric Department.

It will be studied if such video triage is safe and if the patients don't get under-triaged, as well as studying the operators' and parents' experiences of the video call, regarding safety and degree of worry. The project thus aims at improving the triage with new technology, with better patient courses as a result, so that patients without the need for urgent medical assessment and treatment safely can stay at home, and patients with urgent medical attention are directly referred to the hospital. All in all, video triage can thereby reduce the strain on the sick child, its parents and the health services. To the knowledge of the authors, there are no other studies of the effect of video calls in the initial triage of children, and therefore this project will contribute with new knowledge in this area.

Method Project setup A small group of operators, all nurses, has been trained in video triage as part of the above-mentioned project on children with respiratory symptoms. They will offer video calls every other day they are at work, i.e. one-day video triage and the next day regular telephone triage, and so on. During the project period, more operators will be taught in video triage, so that more operators can participate. There will thus be a step-by-step inclusion of operators who carry out video triage. The project thus has the character of a stepped wedge randomized trial.

The results of video days will be compared to results from non-video days. The control group will thus be patients from non-video days.

Patient population: The effect of video triage will be studied on young children with fever, as this patient group is large and frequently contact 1813, and it is expected that the assessment of the general state of these children by video calls is better than by phone calls.

Method of video triage On video days, the operators will offer video calls to anyone who meets the inclusion criteria.

The parents will receive a link on their smartphone, which upon activation starts a video conversation with the operator at 1813. The operator will use the medical history and the video, i.e. both pictures and sound, to make a plan for the child, together with the parent. Apart from the video conversation, the operator has all the normal possibilities as in not-project calls. For example, there is a call-back option, where the operator can call back to the parents after a few hours to hear how the child is after paracetamol administration, amongst other possibilities.

Immediately after the call, the parents will receive an SMS with a link to a questionnaire. They will for example be asked how confident they feel about the assessment of the child; how safe they feel about the plan laid out for the child and what their DOW was before and after the call to 1813. All parents will get a reminder about the questionnaire by SMS 24-48 hours after the call.

After the interview, the operators at 1813 will answer a questionnaire as well. They will be asked about how it was to have additional information about the child's condition by watching and hearing the child on video and how worried they were for the child, among other questions.

On non-video days, the project operators will include similar children for the telephone group . Correspondingly, these parents will also receive an SMS with a link to a questionnaire about their experience of the conversation, and a reminder to respond. As with video days, the operators will have the possibility to use options as in calls that are not part of a project, i.e. for example the possibility of call-back and that parents can send pictures if the operator finds it relevant. It will be noted when these options are being used.

Within 2 to 8 business days after the call, the doctors in the project group will read all enrolled children's hospital reports in the hospitals' electronic records system, to investigate if the children have been at a Pediatric Department within 8 or 48 hours after the 1813 call. If a child has been at the hospital, it will be noted if it was seen at a pediatric urgent care clinic or at the PED, time and diagnosis, temperature measured in hospital, optimally including how temperature was measured, if the child was admitted to the pediatric ward, and if so, for how many days. It will also be registered what kind of paraclinical testing and treatment the child received, if the child was transferred to an intensive care unit, or at worst, got lasting injuries or death.

The data department at the Emergency Services will daily identify the children involved in the project, in that the operators mark the calls in the 1813 record system. The data sheet will include call date and time, symptom code and disposition, i.e. what the child was referred to. The data sheet will also include the calls that have met the inclusion criteria, but where the parent did not want to participate.

Technical set-up for video calling The video solution is provided by GoodSAM Instant-on-Scene, which is already used in several locations in Australia and in the UK and can be used on Apple, Windows and Android phones (https://www.goodsamapp.org/instantOnScene).

Sample size In 2018, there were 177,000 calls concerning children under the age of 6. Of the 177,000, 9% were referred to admission at a Pediatric Department, 30% were referred to a pediatric urgency care clinic, 31% were counseled about self-care and 25% were recommended to contact their GP the next working day, i.e. that 56% stayed at home the day the parents called 1813.

It will be investigated if video triage can result in 10% more parents staying at home with the child in the next 8 hours after the call, i.e. an increase from 56% to 66%. With a power of 80% and two-sided significance of 95%, 774 children divided into two groups should be included, according to openepi (http://www.openepi.com/SampleSize/SSCohort.htm).

The project will be tested for a maximum of 6 months.

Statistical calculations Non-parametric statistics, double-sided and with significance at p-value <0.05.

Possible yield After the completion of the project, the project group expect to know if video calls is an effective new technique that optimizes the triage process, so that more slightly ill children can stay at home the day their parents call 1813. That would be a benefit for the sick child, its parents and a significant socio-economic gain. It will also be known if more severely ill children are referred directly to a Pediatric Emergency Department to a greater extent than today, rather than to an initial assessment in a pediatric urgency care clinic or being referred to staying at home.

At the end of the project, the management of the Copenhagen Emergency Medical Services can use the project's results to decide if video calls should be a permanent option when contacting the Medical Helpline 1813.

It is expected that video triage will support the health services' work to create the most appropriate courses for the children and their families, while at the same time reducing resource consumption.

ELIGIBILITY:
Inclusion Criteria:

* Parents state that the child has fever.
* Parents are calling from a smartphone with Apple, Windows or Android operating system.

Exclusion Criteria:

* The child has already participated.
* The parent does not call from a Danish telephone number.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 801 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Disposition | Disposition is registered by the operator immediately after the call for all patients included, throughout the project period..
  Difference between the arms in the percentage of children that stays at home the first 8 hours after the call, i.e. referral to self-care or GP.

SECONDARY OUTCOMES:
Admittance | The hospital chart of all children is read within 2-8 days after the call for all patients included, throughout the project period.
  Difference between the arms in the percentage of children that is admitted directly to a pediatric emergency department
Hospital visits | The hospital chart of all children is read within 2-8 days after the call for all patients included, throughout the project period..
  Difference between the two arms in how many children that were seen at a hospital at 8 and 48 hours after the call. Also, what temperature did they have, what diagnoses did they receive, were they admitted, and if so for how long, were any children transferred to ICU, and did any children die?
Treatment | The hospital chart of all children is read within 2-8 days after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how many children that received treatment or paraclinical tests, or got a prescription.
Operators: satisfaction | The operators fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how many operators that were satisfied with the call to an acceptable extent or better.
Operators: DOW | The operators fill out a survey immediately after the call for all patients included, throughout the project period..
  Presentation of the DOW in the two groups, and if there are any differences.
Operators: safety | The operators fill out a survey immediately after the call for all patients included, throughout the project period..
  How many operators state that they feel more safe about the disposition choice when having seen the child on video.
Parents: satisfaction with the contact to 1813 | The parents fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how many parents that were satisfied with the contact to 1813 to an acceptable extent or better.
Parents: Questions getting answered | The parents fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how many parents that felt that they got answers to their questions during the call to 1813 to an acceptable extent or better.
Parents: satisfaction about assessment | The parents fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how many parents that felt safe about the assessment of their child to an acceptable extent or better.
Parents: satisfaction about the plan | The parents fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how many parents that felt safe about the plan laid out for their child to an acceptable extent or better.
Parents: DOW before call | The parents fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how they grade their worry BEFORE having talked to the operator at 1813.
Parents: DOW after call | The parents fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how they grade their worry AFTER having talked to the operator at 1813.
Parents: video as a permanent options | The parents fill out a survey immediately after the call for all patients included, throughout the project period..
  The difference in percentage between the two arms in how many that think that video should be made a permanent option at 1813
Economical consequences | Can be calculated when the project no longer enrolls children, the inclusion is expected to be ready after approximately 4 months.
  Calculation of how many visits at the hospital that could be avoided because of video triage.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Cortes, M.D., Study Chair — Department of Pediatrics, Copenhagen University Hopsital Hvidovre
Locations (1):
- Emergency Medical Services, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen MV. Data, controlling and IT section, Copenhagen Emergency Services. January 2019.
- [Background] Boisen AS. Implementeringen af Enstrenget og Visiteret Akutsystem i Region Hovedstaden - en analyse af samspillet mellem organisatorisk forandring og brugeradfærd. Institut for Folkesundhedsvidenskab, Københavns Universitet; 2015
- [Background] Børns brug af regionale sundhedsydelser. Center for Sundhed - Enhed for Tværsektoriel Udvikling. Region Hovedstaden. 2017. https://www.regionh.dk/til-fagfolk/Sundhed/Tvaersektorielt-samarbejde/samarbejdspulje-og-forebyggelse/Documents/rapport-boerns-brug-regionale-sundhedsydelser.pdf
- [Background] Analyse af børns brug af sundhedsydelser. Center for Sundhed - Enhed for Tværsektoriel Udvikling. Region Hovedstaden. 2017. https://www.regionh.dk/til-fagfolk/Sundhed/Tvaersektorielt-samarbejde/samarbejdspulje-og-forebyggelse/Documents/analyse_af_boerns_brug_af_sundhedsydelser.pdf
- [Background] Nijman RG, Oostenbrink R, Dons EM, Bouwhuis CB, Moll HA. Parental fever attitude and management: influence of parental ethnicity and child's age. Pediatr Emerg Care. 2010 May;26(5):339-42. doi: 10.1097/PEC.0b013e3181db1dce. PMID 20404784
- [Background] Kelly M, Sahm LJ, Shiely F, O'Sullivan R, McGillicuddy A, McCarthy S. Parental knowledge, attitudes and beliefs regarding fever in children: an interview study. BMC Public Health. 2016 Jul 11;16:540. doi: 10.1186/s12889-016-3224-5. PMID 27401677
- [Background] Crocetti M, Moghbeli N, Serwint J. Fever phobia revisited: have parental misconceptions about fever changed in 20 years? Pediatrics. 2001 Jun;107(6):1241-6. doi: 10.1542/peds.107.6.1241. PMID 11389237
- [Background] Parkinson GW, Gordon KE, Camfield CS, Fitzpatrick EA. Anxiety in parents of young febrile children in a pediatric emergency department: why is it elevated? Clin Pediatr (Phila). 1999 Apr;38(4):219-26. doi: 10.1177/000992289903800403. PMID 10326177
- [Background] Lægehåndbogen. Feber hos børn. https://www.sundhed.dk/sundhedsfaglig/laegehaandbogen/paediatri/symptomer-og-tegn/feber-hos-boern/
- [Background] Pantell RH, Newman TB, Bernzweig J, Bergman DA, Takayama JI, Segal M, Finch SA, Wasserman RC. Management and outcomes of care of fever in early infancy. JAMA. 2004 Mar 10;291(10):1203-12. doi: 10.1001/jama.291.10.1203. PMID 15010441
- [Background] Woll C, Neuman MI, Aronson PL. Management of the Febrile Young Infant: Update for the 21st Century. Pediatr Emerg Care. 2017 Nov;33(11):748-753. doi: 10.1097/PEC.0000000000001303. PMID 29095773
- [Background] Van den Bruel A, Aertgeerts B, Bruyninckx R, Aerts M, Buntinx F. Signs and symptoms for diagnosis of serious infections in children: a prospective study in primary care. Br J Gen Pract. 2007 Jul;57(540):538-46. PMID 17727746
- [Background] Verbakel JY, Van den Bruel A, Thompson M, Stevens R, Aertgeerts B, Oostenbrink R, Moll HA, Berger MY, Lakhanpaul M, Mant D, Buntinx F; European Research Network on Recognising Serious Infection (ERNIE). How well do clinical prediction rules perform in identifying serious infections in acutely ill children across an international network of ambulatory care datasets? BMC Med. 2013 Jan 15;11:10. doi: 10.1186/1741-7015-11-10. PMID 23320738
- [Background] Van den Bruel A, Bartholomeeusen S, Aertgeerts B, Truyers C, Buntinx F. Serious infections in children: an incidence study in family practice. BMC Fam Pract. 2006 Mar 28;7:23. doi: 10.1186/1471-2296-7-23. PMID 16569232
- [Background] Kool M, Elshout G, Moll HA, Koes BW, van der Wouden JC, Berger MY. Duration of fever and course of symptoms in young febrile children presenting with uncomplicated illness. J Am Board Fam Med. 2013 Jul-Aug;26(4):445-52. doi: 10.3122/jabfm.2013.04.120265. PMID 23833160
- [Background] Gamst-Jensen H, Huibers L, Pedersen K, Christensen EF, Ersboll AK, Lippert FK, Egerod I. Self-rated worry in acute care telephone triage: a mixed-methods study. Br J Gen Pract. 2018 Mar;68(668):e197-e203. doi: 10.3399/bjgp18X695021. Epub 2018 Feb 12. PMID 29440015
- [Background] Gamst-Jensen H. Patients' self-assessment of illness and injury in telephone triage using a novel degree-of-worry scale. Ph.D. dissertation. Faculty of Health and Medical Science, University of Copenhagen; 2018.
- [Background] Olson CA, Thomas JF. Telehealth: No Longer an Idea for the Future. Adv Pediatr. 2017 Aug;64(1):347-370. doi: 10.1016/j.yapd.2017.03.009. No abstract available. PMID 28688597
- [Background] COMMITTEE ON PEDIATRIC WORKFORCE; Marcin JP, Rimsza ME, Moskowitz WB. The Use of Telemedicine to Address Access and Physician Workforce Shortages. Pediatrics. 2015 Jul;136(1):202-9. doi: 10.1542/peds.2015-1253. PMID 26122802
- [Background] Regioner på vej med ny app: Hver tredje konsultation kan ske online. Dagens Medicin. 2018. https://dagensmedicin.dk/danske-regioner-lancerer-ny-app-hver-tredje-konsultation-kan-ske-online/
- [Background] Videokonsultationer skal få praktiserende læger til Mors og til andre lægedækningstruede områder. Region Nordjylland. http://rn.dk/service/nyhedsliste-rn/nyhed?id=48723d23-88da-4759-a685-9c9336bc6093
- [Background] Ekeland AG, Bowes A, Flottorp S. Effectiveness of telemedicine: a systematic review of reviews. Int J Med Inform. 2010 Nov;79(11):736-71. doi: 10.1016/j.ijmedinf.2010.08.006. PMID 20884286
- [Background] Siew L, Hsiao A, McCarthy P, Agarwal A, Lee E, Chen L. Reliability of Telemedicine in the Assessment of Seriously Ill Children. Pediatrics. 2016 Mar;137(3):e20150712. doi: 10.1542/peds.2015-0712. Epub 2016 Feb 5. PMID 26908666
- [Background] McCarthy PL, Sharpe MR, Spiesel SZ, Dolan TF, Forsyth BW, DeWitt TG, Fink HD, Baron MA, Cicchetti DV. Observation scales to identify serious illness in febrile children. Pediatrics. 1982 Nov;70(5):802-9. No abstract available. PMID 7133831
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Derived] Gren C, Hasselager AB, Linderoth G, Frederiksen MS, Folke F, Ersboll AK, Gamst-Jensen H, Cortes D. Video triage in calls concerning children with fever at an out-of-hours medical helpline: a prospective quality improvement study. Scand J Trauma Resusc Emerg Med. 2023 Aug 29;31(1):41. doi: 10.1186/s13049-023-01106-9. PMID 37644510